CLINICAL TRIAL: NCT05163249
Title: A Prospective, Pilot Study of First-line Osimertinib With or Without Savolitinib in de Novo MET Positive, EGFR-mutant NSCLCs (FLOWERS)
Brief Title: Osimertinib With or Without Savolitinib as 1L in de Novo MET+, EGFR+ NSCLC
Acronym: FLOWERS
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Guangdong Association of Clinical Trials (Other)
Responsible Party: Principal Investigator, Jin-Ji Yang, Principal Investigator, Guangdong Association of Clinical Trials
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CTONG 2008
Record Dates: First submitted 2021-12-06; First posted 2021-12-20 (Actual); Last update posted 2024-02-09 (Actual); Status verified 2024-02

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: non-small-cell lung cancer; Epidermal growth factor receptor; de novo MET amplification; Targeted Therapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — osimertinib; 1-(1-(imidazo(1,2-a)pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-(1,2,3)triazolo(4,5-b)pyrazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1: osimertinib, 80mg, daily, P.O. (Active Comparator): Patients will continue to receive study medication in 28 day cycles until objective disease progression, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criterion is met.
  Patients who progress on first-line treatment of osimertinib monotherapy will have the opportunity to receive second-line treatment of osimertinib plus savolitinib after confirmation of MET status at disease progression.
  Interventions: Drug: Osimertinib
- Cohort 2: osimertinib 80mg daily, P.O. and savolitinib 300mg BID, P.O. (Experimental): All eligible patients will be randomized to receive treatment with osimertinib (80 mg daily) or osimertinib (80 mg daily) in combination with savolitinib (300 mg BID) in this study. Treatment will continue until either objective disease progression, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criterion is met.
  Patients in Cohort 2 can continue on savolitinib monotherapy (if osimertinib was stopped earlier) or osimertinib monotherapy (if savolitinib was stopped earlier) until objective disease progression or meet any of the discontinuation criteria.
  Interventions: Drug: Osimertinib; Drug: Savolitinib

INTERVENTIONS:
Drug: Osimertinib — osimertinib, 80mg, daily, P.O. Until objective disease progression, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criteria is met
  Other Names: AZD9291
Drug: Savolitinib — savolitinib 300mg BID, P.O. Until objective disease progression, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criteria is met
  Other Names: HMPL-504
  Arms: Cohort 2: osimertinib 80mg daily, P.O. and savolitinib 300mg BID, P.O.

SUMMARY:
This is a prospective, pilot, two-arm, randomized, multicenter study exploring the efficacy and safety of osimertinib with or without savolitinib as first-line therapy in patients with de novo MET positive, EGFR-mutant advanced NSCLC.

DETAILED DESCRIPTION:
Approximately 44 eligible patients will be enrolled to randomly assigned to study interventions so that approximately 40 evaluable participants complete the study, based on an assumption of 10% of participants not completing the study.

All eligible patients will be randomized in a 1:1 ratio to receive treatment with osimertinib (80 mg daily) or osimertinib (80 mg daily) in combination with savolitinib (300 mg BID) in this study. Treatment will continue until either objective disease progression, unacceptable toxicity occurs, consent is withdrawn or another discontinuation criterion is met.

Patients who progress on first-line treatment of osimertinib monotherapy will have the opportunity to receive second-line treatment of osimertinib plus savolitinib after confirmation of MET status at disease progression.

ELIGIBILITY:
Inclusion Criteria:

Participants are eligible to be included in the study only if all of the following criteria apply:

Informed consent

1. Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol.
2. Provision of signed and dated, written ICF prior to any mandatory study specific procedures, sampling, and analyses.

   Age
3. Participant must be ≥18 years at the time of signing the ICF. All genders are permitted.

   Type of Participant and Disease Characteristics
4. Histologically or cytologically confirmed locally advanced or metastatic EGFRm+ NSCLC harbouring an EGFR mutation known to be associated with EGFR TKI sensitivity.
5. Has not received any systemic treatment of advanced NSCLC.

   * Prior adjuvant/neo-adjuvant therapy completed > 6 months before screening is allowed.
6. MET amplification/high expression as determined by FISH, IHC or NGS testing on tumor tissue collected before any systemic treatment in first line.

   * MET high expression by IHC, 3+ in ≥75% of tumor cells
   * increased MET gene copy number by FISH, MET gene copy ≥5 or MET / CEP7 ratio ≥2; or by tissue NGS, ≥20% tumour cells, ≥200x sequencing depth of coverage and CN ≥5.
   * Local IHC, FISH and pre-existing local NGS results are acceptable, central FISH and central NGS confirmation is highly suggested if tissue sample available.
7. WHO or Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 with no deterioration over the previous 2 weeks prior to baseline or day of first dosing and a minimum life expectancy of 12 weeks.
8. At least 1 lesion that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) or magnetic resonance imaging (MRI) and is suitable for accurate repeated measurements.
9. Adequate haematological function defined as:

   * Haemoglobin≥8.5 g/dL (no transfusion in the past 2 weeks).
   * Absolute neutrophil count ≥1.5×109/L.
   * Platelet count ≥100,000/μL (no transfusion in the past 10 days)
10. Adequate liver function defined as:

    * Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 x the upper limit of normal (ULN) with total bilirubin (TBL) ≤ ULN
    * OR TBL >ULN to ≤1.5x ULN with ALT and AST ≤ ULN
11. Adequate renal function defined as a creatinine <1.5 times the institutional ULN OR a glomerular filtration rate ≥50 mL/min, as assessed using the standard methodology at the investigating centre (eg, Cockcroft-Gault, Modification of Diet in Renal Disease or Chronic Kidney Disease Epidemiology Collaboration formulae, ethylenediaminetetraacetic acid clearance or 24-hour urine collection). Confirmation of creatinine clearance is only required when creatinine is >1.5 times ULN.
12. Adequate coagulation parameters, defined as:

    * International Normalisation Ratio (INR) <1.5 x ULN and activated partial thromboplastin time <1.5 x ULN unless patients are receiving therapeutic anti coagulation which affects these parameters.
13. Patients with known tumor thrombus or deep vein thrombosis are eligible if clinically stable on low molecular weight heparin (LMWH) for ≥2 weeks.
14. Ability to swallow and retain oral medications.
15. Willingness and ability to comply with study and follow-up procedures.

    Reproduction
16. Females must be using highly effective contraceptive measures (see Section 5.3.2), and have a negative pregnancy test (serum) for women of childbearing potential, or must have evidence of non-childbearing potential by fulfilling one of the following criteria at screening:

    * Post-menopausal is defined as aged more than 50 years and amenorrhoeic for at least 12 months following cessation of all exogenous hormonal treatments.
    * Women under the age of 50 years would be considered postmenopausal if they have been amenorrhoeic for 12 months or more following cessation of exogenous hormonal treatments and with luteinizing hormone and follicle stimulating hormone levels in the post-menopausal range for the institution.
    * Women with documentation of irreversible surgical sterilisation by hysterectomy, bilateral oophorectomy or bilateral salpingectomy but not tubal ligation.
    * Further information is available in Appendix F (Contraception Requirements).
17. Male patients with a female partner of childbearing potential should be willing to use barrier contraception during the study and for 6 months following discontinuation of study drug. Patients should refrain from donating sperm from the start of dosing until 6 months after discontinuing study treatment.

Exclusion Criteria:

Participants are excluded from the study if any of the following criteria apply:

Medical Conditions

1. As judged by the investigator, active gastrointestinal disease or other condition that will interfere significantly with the absorption, distribution, metabolism, or excretion of oral therapy (eg, ulcerative disease, uncontrolled nausea, vomiting, diarrhoea Grade ≥2, malabsorption syndrome or previous significant bowel resection).
2. Any of the following cardiac diseases currently or within the last 6 months:

   * Unstable angina pectoris
   * Congestive heart failure (New York Heart Association [NYHA] ≥Grade 2)
   * Acute myocardial infarction
   * Stroke or transient ischemic attack
   * Uncontrolled hypertension (BP ≥150/95 mmHg despite medical therapy).
   * Mean resting correct QT interval (QTcF) >470 msec for women and >450 msec for men at Screening, obtained from 3 ECGs using the screening clinic ECG machine derived QTcF value.
   * Any factors that may increase the risk of QTcF prolongation or risk of arrhythmic events such as heart failure, electrolyte abnormalities (including: Serum/plasma potassium < LLN; Serum/plasma magnesium < LLN; Serum/plasma calcium < LLN), congenital or familial long QT syndrome, family history of unexplained sudden death under 40 years of age in first-degree relatives or any concomitant medication known to prolong the QT interval and cause Torsade de Pointes.
   * Any clinically important abnormalities in rhythm, conduction or morphology of resting ECGs, eg, complete left bundle branch block, third degree heart block, second degree heart block, P-R interval >250 msec.
   * Acute coronary syndrome
3. Wide field radiotherapy (including therapeutic radioisotopes such as strontium 89) administered ≤28 days or limited field radiation for palliation ≤7 days prior to starting study drug or has not recovered from side effects of such therapy.
4. Major surgical procedures ≤28 days of beginning study drug or minor surgical procedures ≤7 days. No waiting is required following port-a-cath placement.
5. As judged by the investigator, any evidence of severe or uncontrolled systemic diseases, including renal transplant, active bleeding diatheses or uncontrolled hypertension, which in the investigator's opinion makes it undesirable for the patient to participate in the trial or which would jeopardise compliance with the protocol.
6. Active hepatitis B (HBV) (positive HBV surface antigen [HBsAg] result) or hepatitis C (HCV). Viral testing is not required for assessment of eligibility for the study. Patients with a past or resolved HBV or HCV infection are eligible if:

   * Negative for HBsAg and positive for hepatitis B core antibody [anti-HBc] or
   * Positive for HBsAg, but for >6 months have had normal transaminases and HBV DNA levels between 0 to 2000 IU/mL (inactive carrier state) and willing to start and maintain antiviral treatment for at least the duration of the study.
   * HBV DNA levels >2000 IU/mL but on prophylactic antiviral treatment for the past 3 months and will maintain the antiviral treatment during the study.
   * Patients with positive HCV antibody are eligible only if the polymerase chain reaction is negative for HCV ribonucleic acid.
7. Presence of other active cancers, or history of treatment for invasive cancer, within the last 5 years. Patients with Stage I cancer who have received definitive local treatment at least 3 years previously, and are considered unlikely to recur are eligible. All patients with previously treated in situ carcinoma (ie, non-invasive) are eligible, as are patients with history of non-melanoma skin cancer.
8. Unresolved toxicities from any prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment/randomization with the exception of alopecia
9. Spinal cord compression or brain metastases unless asymptomatic, stable, and not requiring steroids for at least 2 weeks prior to start of study intervention. Subjects with leptomeningeal metastases are ineligible.
10. Past medical history of ILD/pneumonitis, drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active ILD.
11. Known serious active infection including, but not limited to, tuberculosis, or human immunodeficiency virus (positive human immunodeficiency virus 1/2 antibodies). Testing is not required for assessment of eligibility for the study..
12. Known history of liver fibrosis/cirrhosis.
13. Known contraindications to osimertinib administration.
14. Known hypersensitivity to the active or inactive excipients of osimertinib or savolitinib or drugs with a similar chemical structure or class.

    Prior/Concomitant Therapy
15. Prior exposure to HGF/MET inhibitors, e.g., foretinib, crizotinib, cabozantinib, merestinib, onartuzumab, capmatinib, tepotinib, etc..
16. Prior exposure to EGFR TKI.
17. Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be strong inducers of CYP3A4, strong inhibitors of CYP1A2, within 2 weeks of the first dose of study treatment (3 weeks for St John's Wort) will be excluded. All patients must try to avoid concomitant use of any medications, herbal supplements and/or ingestion of foods with known inducer effects on CYP3A4 during the study and for 3 months later the last dose intake.

    Prior/Concurrent Clinical Study Experience
18. Participation in another clinical study with a study interventional medication administered within five half-lives of the compound or 3 months, whichever is greater or investigational medicinal device administered in the last 30 days prior to randomisation/first dose of study intervention or concurrent enrolment in another clinical study, unless it is an observational (non interventional) clinical study or during the follow-up period of an interventional study.

    Other Exclusions
19. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca staff and/or staff at the study site).
20. Judgment by the investigator that the participant should not participate in the study if the participant is unlikely to comply with study procedures, restrictions and requirements.
21. For women only-Currently breastfeeding.
22. Previous enrolment in the present study.
23. Without civil capacity or with restricted civil capacity.
24. Any other reasons judged by the leading investigator to prevent the subject from participating in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2022-05-31 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
ORR | 12 weeks after the last patient enrolled
  Objective response rate (ORR) of the tumor using Investigator assessment as defined by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1)

SECONDARY OUTCOMES:
PFS | 18 months after the last patient enrolled
  Progression-free survival (Investigator assessment as defined by RECIST 1.1)
DoR | 18 months after the last patient enrolled
  The duration between the date the criteria for complete response or partial response was first measured (first record shall prevail) and the date of disease recurrence or progression as objectively recorded
DCR | 18 months after the last patient enrolled
  the incidence of complete response, partial response and stable disease
percentage change from baseline in tumor size | 12 weeks after the last patient enrolled
  Absolute change and percentage change from baseline in TL's tumor size at 12 weeks will be based on RECIST TLs measurements taken at baseline and at Week 12
OS | 18 months after the last patient enrolled
  Overall survival (OS) is defined as the time from the start of treatment until death due to any cause
12m OS rate by Investigator assessment | 12 months after the last patient enrolled
  Proportion alive at 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Ji Yang, MD, Principal Investigator — Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences
Locations (1):
- Guangdong Lung Cancer Institute, Guangdong General Hospital, Guangdong Academy of Medical Sciences, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blakely CM, Watkins TBK, Wu W, Gini B, Chabon JJ, McCoach CE, McGranahan N, Wilson GA, Birkbak NJ, Olivas VR, Rotow J, Maynard A, Wang V, Gubens MA, Banks KC, Lanman RB, Caulin AF, St John J, Cordero AR, Giannikopoulos P, Simmons AD, Mack PC, Gandara DR, Husain H, Doebele RC, Riess JW, Diehn M, Swanton C, Bivona TG. Evolution and clinical impact of co-occurring genetic alterations in advanced-stage EGFR-mutant lung cancers. Nat Genet. 2017 Dec;49(12):1693-1704. doi: 10.1038/ng.3990. Epub 2017 Nov 6. PMID 29106415
- [Background] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Background] Chen W, Zheng R, Baade PD, Zhang S, Zeng H, Bray F, Jemal A, Yu XQ, He J. Cancer statistics in China, 2015. CA Cancer J Clin. 2016 Mar-Apr;66(2):115-32. doi: 10.3322/caac.21338. Epub 2016 Jan 25. PMID 26808342
- [Background] Choueiri TK, Halabi S, Sanford BL, Hahn O, Michaelson MD, Walsh MK, Feldman DR, Olencki T, Picus J, Small EJ, Dakhil S, George DJ, Morris MJ. Cabozantinib Versus Sunitinib As Initial Targeted Therapy for Patients With Metastatic Renal Cell Carcinoma of Poor or Intermediate Risk: The Alliance A031203 CABOSUN Trial. J Clin Oncol. 2017 Feb 20;35(6):591-597. doi: 10.1200/JCO.2016.70.7398. Epub 2016 Nov 14. PMID 28199818
- [Background] Duan J, Xu J, Wang Z, Bai H, Cheng Y, An T, Gao H, Wang K, Zhou Q, Hu Y, Song Y, Ding C, Peng F, Liang L, Hu Y, Huang C, Zhou C, Shi Y, Han J, Wang D, Tian Y, Yang Z, Zhang L, Chuai S, Ye J, Zhu G, Zhao J, Wu YL, Wang J. Refined Stratification Based on Baseline Concomitant Mutations and Longitudinal Circulating Tumor DNA Monitoring in Advanced EGFR-Mutant Lung Adenocarcinoma Under Gefitinib Treatment. J Thorac Oncol. 2020 Dec;15(12):1857-1870. doi: 10.1016/j.jtho.2020.08.020. Epub 2020 Sep 9. PMID 32916309
- [Background] Gainor JF, Niederst MJ, Lennerz JK, Dagogo-Jack I, Stevens S, Shaw AT, Sequist LV, Engelman JA. Dramatic Response to Combination Erlotinib and Crizotinib in a Patient with Advanced, EGFR-Mutant Lung Cancer Harboring De Novo MET Amplification. J Thorac Oncol. 2016 Jul;11(7):e83-5. doi: 10.1016/j.jtho.2016.02.021. Epub 2016 Mar 14. No abstract available. PMID 26988570
- [Background] Hong S, Gao F, Fu S, Wang Y, Fang W, Huang Y, Zhang L. Concomitant Genetic Alterations With Response to Treatment and Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors in Patients With EGFR-Mutant Advanced Non-Small Cell Lung Cancer. JAMA Oncol. 2018 May 1;4(5):739-742. doi: 10.1001/jamaoncol.2018.0049. PMID 29596544
- [Background] Jia H, Dai G, Weng J, Zhang Z, Wang Q, Zhou F, Jiao L, Cui Y, Ren Y, Fan S, Zhou J, Qing W, Gu Y, Wang J, Sai Y, Su W. Discovery of (S)-1-(1-(Imidazo[1,2-a]pyridin-6-yl)ethyl)-6-(1-methyl-1H-pyrazol-4-yl)-1H-[1,2,3]triazolo[4,5-b]pyrazine (volitinib) as a highly potent and selective mesenchymal-epithelial transition factor (c-Met) inhibitor in clinical development for treatment of cancer. J Med Chem. 2014 Sep 25;57(18):7577-89. doi: 10.1021/jm500510f. Epub 2014 Sep 15. PMID 25148209
- [Background] Lai GGY, Lim TH, Lim J, Liew PJR, Kwang XL, Nahar R, Aung ZW, Takano A, Lee YY, Lau DPX, Tan GS, Tan SH, Tan WL, Ang MK, Toh CK, Tan BS, Devanand A, Too CW, Gogna A, Ong BH, Koh TPT, Kanesvaran R, Ng QS, Jain A, Rajasekaran T, Yuan J, Lim TKH, Lim AST, Hillmer AM, Lim WT, Iyer NG, Tam WL, Zhai W, Tan EH, Tan DSW. Clonal MET Amplification as a Determinant of Tyrosine Kinase Inhibitor Resistance in Epidermal Growth Factor Receptor-Mutant Non-Small-Cell Lung Cancer. J Clin Oncol. 2019 Apr 10;37(11):876-884. doi: 10.1200/JCO.18.00177. Epub 2019 Jan 24. PMID 30676858
- [Background] Masters GA, Temin S, Azzoli CG, Giaccone G, Baker S Jr, Brahmer JR, Ellis PM, Gajra A, Rackear N, Schiller JH, Smith TJ, Strawn JR, Trent D, Johnson DH; American Society of Clinical Oncology Clinical Practice. Systemic Therapy for Stage IV Non-Small-Cell Lung Cancer: American Society of Clinical Oncology Clinical Practice Guideline Update. J Clin Oncol. 2015 Oct 20;33(30):3488-515. doi: 10.1200/JCO.2015.62.1342. Epub 2015 Aug 31. PMID 26324367
- [Background] Pisters KM, Le Chevalier T. Adjuvant chemotherapy in completely resected non-small-cell lung cancer. J Clin Oncol. 2005 May 10;23(14):3270-8. doi: 10.1200/JCO.2005.11.478. PMID 15886314
- [Background] Reck M, Popat S, Reinmuth N, De Ruysscher D, Kerr KM, Peters S; ESMO Guidelines Working Group. Metastatic non-small-cell lung cancer (NSCLC): ESMO Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2014 Sep;25 Suppl 3:iii27-39. doi: 10.1093/annonc/mdu199. Epub 2014 Aug 11. No abstract available. PMID 25115305
- [Background] Sequist LV, Han JY, Ahn MJ, Cho BC, Yu H, Kim SW, Yang JC, Lee JS, Su WC, Kowalski D, Orlov S, Cantarini M, Verheijen RB, Mellemgaard A, Ottesen L, Frewer P, Ou X, Oxnard G. Osimertinib plus savolitinib in patients with EGFR mutation-positive, MET-amplified, non-small-cell lung cancer after progression on EGFR tyrosine kinase inhibitors: interim results from a multicentre, open-label, phase 1b study. Lancet Oncol. 2020 Mar;21(3):373-386. doi: 10.1016/S1470-2045(19)30785-5. Epub 2020 Feb 3. PMID 32027846
- [Background] Shi Y, Au JS, Thongprasert S, Srinivasan S, Tsai CM, Khoa MT, Heeroma K, Itoh Y, Cornelio G, Yang PC. A prospective, molecular epidemiology study of EGFR mutations in Asian patients with advanced non-small-cell lung cancer of adenocarcinoma histology (PIONEER). J Thorac Oncol. 2014 Feb;9(2):154-62. doi: 10.1097/JTO.0000000000000033. PMID 24419411
- [Background] Soria JC, Wu YL, Nakagawa K, Kim SW, Yang JJ, Ahn MJ, Wang J, Yang JC, Lu Y, Atagi S, Ponce S, Lee DH, Liu Y, Yoh K, Zhou JY, Shi X, Webster A, Jiang H, Mok TS. Gefitinib plus chemotherapy versus placebo plus chemotherapy in EGFR-mutation-positive non-small-cell lung cancer after progression on first-line gefitinib (IMPRESS): a phase 3 randomised trial. Lancet Oncol. 2015 Aug;16(8):990-8. doi: 10.1016/S1470-2045(15)00121-7. Epub 2015 Jul 6. PMID 26159065
- [Background] Wang F, Diao XY, Zhang X, Shao Q, Feng YF, An X, Wang HY. Identification of genetic alterations associated with primary resistance to EGFR-TKIs in advanced non-small-cell lung cancer patients with EGFR sensitive mutations. Cancer Commun (Lond). 2019 Mar 2;39(1):7. doi: 10.1186/s40880-019-0354-z. PMID 30823937
- [Background] Wang Z, Cheng Y, An T, Gao H, Wang K, Zhou Q, Hu Y, Song Y, Ding C, Peng F, Liang L, Hu Y, Huang C, Zhou C, Shi Y, Zhang L, Ye X, Zhang M, Chuai S, Zhu G, Hu J, Wu YL, Wang J. Detection of EGFR mutations in plasma circulating tumour DNA as a selection criterion for first-line gefitinib treatment in patients with advanced lung adenocarcinoma (BENEFIT): a phase 2, single-arm, multicentre clinical trial. Lancet Respir Med. 2018 Sep;6(9):681-690. doi: 10.1016/S2213-2600(18)30264-9. Epub 2018 Jul 17. PMID 30017884
- [Background] Yu HA, Suzawa K, Jordan E, Zehir A, Ni A, Kim R, Kris MG, Hellmann MD, Li BT, Somwar R, Solit DB, Berger MF, Arcila M, Riely GJ, Ladanyi M. Concurrent Alterations in EGFR-Mutant Lung Cancers Associated with Resistance to EGFR Kinase Inhibitors and Characterization of MTOR as a Mediator of Resistance. Clin Cancer Res. 2018 Jul 1;24(13):3108-3118. doi: 10.1158/1078-0432.CCR-17-2961. Epub 2018 Mar 12. PMID 29530932
- [Derived] Li A, Feng WN, Li J, Xu BF, Zhao J, Jia Y, Tang KJ, Li YS, Zhou CZ, Fan Y, Xu CR, Sun YL, Chen HJ, Yan HH, Shi ZK, Yang JJ. Osimertinib with or without savolitinib as first-line treatment for MET-aberrant, EGFR-mutant NSCLC: randomized phase 2 trial (FLOWERS). Nat Commun. 2026 Jan 13. doi: 10.1038/s41467-025-67950-8. Online ahead of print. PMID 41530133
- [Derived] Li A, Chen HJ, Yang JJ. Design and Rationale for a Phase II, Randomized, Open-Label, Two-Cohort Multicenter Interventional Study of Osimertinib with or Without Savolitinib in De Novo MET Aberrant, EGFR-Mutant Patients with Advanced Non-Small-Cell Lung Cancer: The FLOWERS Trial. Clin Lung Cancer. 2023 Jan;24(1):82-88. doi: 10.1016/j.cllc.2022.09.009. Epub 2022 Sep 30. PMID 36333268